CLINICAL TRIAL: NCT04841850
Title: Clinic And Biologic Efficiency And Tolerance Of Oral Immunotherapy Protocol In Hazelnut Allergic Children
Brief Title: Efficiency And Tolerance Of Hazelnut Oral Immunotherapy Protocol In Hazelnut Allergic Children
Acronym: ENOIME
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 186
Record Dates: First submitted 2021-04-08; First posted 2021-04-12 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-03

CONDITIONS: Allergy, Nut; Pediatric ALL
Keywords: Hazelnut; Oral Immunotherapy; Children; Protocol; Efficiency; Tolerance
MeSH Terms: conditions — Nut Hypersensitivity; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hazelnut allergic children under oral immunotherapy: * Children Under eighteen years of age
  * Convincing clinical history of hazelnut allergy
  * Positive hazelnut prick test or specific IgE
  * Under IOT hazelnut protocol in pneumology and allergology-paediatric departement of the Mother and Child Hospital in Bron
  Interventions: Other: Clinical and biological characteristics

INTERVENTIONS:
Other: Clinical and biological characteristics — * Age at beginning of IOT
  * Sex
  * Atopic and non atopic Comorbidities
  * Sensitization to aero-allergens
  * Sensitization to trophallergens
  * Stage of severity of the elicited reaction
  * Hazelnut Specific IgE + Cor a 1,8,9,14 before IOT and during follow up
  * Hazelnut skin prick test before IOT and during follow up
  * Adverse effects of IOT and their stage (in hospital and at home)
  * Use of adrenaline auto-injector (in hospital and at home)
  * Maintenance dose

SUMMARY:
Prevalence of food allergy in the world has been inscreasing in recent years. Among nut allergy, hazelnut allergy is the most widespread in Europe and particularly in France. The current treatment for hazelnut allergy is based on eviction and wearing of an emergency kit with adrenaline auto-injector pens, to be used in the event of severe anaphylactic reaction. Oral immunotherapy (OIT) is a treatment that is now increasingly being offered as an alternatice to eviction. There are few published data concerning hazelnut OIT in Europe, where its consumption is nevertheless very high.

The main objective of our study is to evaluate the clinical efficacy of the hazelnut OIT protocol, implemented since 2015 in the pneumology and allergology-paediatric department of the Mother and Child Hospital in Bron, in hazelnut allergic children under 18 years old.

The secondary objectives will be to evaluate the biological efficacy and clinical tolerance of the protocol.

The study is retrospective and observational, and is based on the collection of medical data from patient records.

ELIGIBILITY:
Inclusion Criteria:

* Aged Under eighteen years old
* Hazelnut allergy (clinically and biologically)
* Under IOT hazelnut protocol in Pneumo/allergology-paediatric departement of the Mother and Child hospital in Bron

Exclusion Criteria:

* Lack of consent to be included in the study (by their parents)
* Age > 18 years old

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children aged under eighteen. With hazelnut allergy (convincing clinical history and positivity of hazelnut skin prick test history or specific IgE) Under IOT hazelnut protocol in Pneumology/allergology-paediatric department of the Mother and Child Hospital in Bron
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
the proportion of patients in maintenance phase at the one-year consultation | at the one-year consultation
  Patients are in maintenance phase at the end of the up-dosing phase and take regularly a quantity of hazelnut, usually superior to 800 mg, considered an acceptable protective dose

CONTACTS AND LOCATIONS:
Locations (1):
- Pneumology allergology-paediatric department of the Mother and Child Hospital, Bron, France

REFERENCES:
- [Derived] Sabouraud M, Bierme P, Andre-Gomez SA, Villard-Truc F, Payot F, Correard AK, Garnier L, Braun C. Real-life experience with hazelnut oral immunotherapy. Ann Allergy Asthma Immunol. 2022 Apr;128(4):432-438. doi: 10.1016/j.anai.2022.01.002. Epub 2022 Jan 8. PMID 35007745